CLINICAL TRIAL: NCT01996709
Title: Effectiveness of a Marketed One-Step Peroxide Lens Care Solution in Symptomatic Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A01337
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Refractive Error
Keywords: Silicone hydrogel contact lenses; Multi-purpose solution; Lid Papillae; Palpebral Roughness
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clear Care (Experimental): Hydrogen peroxide-based contact lens solution used with habitual contact lenses for 90 days
  Interventions: Device: Hydrogen peroxide-based contact lens solution; Device: Habitual contact lenses
- Habitual MPS (Active Comparator): Habitual contact lens solution used with habitual contact lenses for 90 days
  Interventions: Device: Habitual contact lens solution; Device: Habitual contact lenses

INTERVENTIONS:
Device: Hydrogen peroxide-based contact lens solution
  Other Names: Clear Care®
  Arms: Clear Care
Device: Habitual contact lens solution — Biguanide-preserved
  Arms: Habitual MPS
Device: Habitual contact lenses — Silicone hydrogel contact lenses with a biweekly or monthly replacement schedule

SUMMARY:
The purpose of this study is to assess improvement of palpebral roughness and associated symptoms with 3 months use of Clear Care®.

ELIGIBILITY:
Inclusion Criteria:

* Current biweekly or monthly silicone hydrogel contact lens wearer (excluding Air Optix® brand) and have worn these lenses bilaterally for at least three (3) months prior to Visit 1 (daily wear use only).
* Symptoms of contact lens discomfort as defined by the protocol.
* Habitual use of a biguanide-preserved multi-purpose solution for at least 30 days prior to Visit 1.
* Mild to severe (grade 2-4) Investigator rated palpebral roughness in one or more zones of either eye.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Extended (over-night) contact lens wearer.
* Any systemic or ocular disease or disorder (refractive disorder allowed and mild dry eye with successful contact lens wear is permitted), complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study.
* Topical ocular over the counter (OTC) or prescribed medications, with the exception of contact lens rewetting drops, within 7 days of enrollment.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Zoota, MPH, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 12 study centers located in the US.
Pre-assignment Details: Of the 142 enrolled, 8 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (134).
Period: Overall Study
Arm/Group | Clear Care | Habitual MPS
Started | 66 | 68
Completed | 61 | 67
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Subject Non-Compliant | 1 | 0
Not completed — Failed Inclusion/Exclusion Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis group includes all subjects who were exposed to a study regimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clear Care | Habitual MPS | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (11.55) | 31.4 (7.65) | 32.2 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 55 | 104
  Male | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Investigator Rated Lid Papillae Maximum Score at Day 90
Description: Lid papillae (bumps on the inner eyelid) were assessed by the investigator using slit-lamp biomicroscopy and classified independently for the four palpebral zones (upper lid=1-3; lower lid=4) on a 5-point forced choice scale, where 0 = None; 1 = Slight (diffuse papillae); 2 = Mild (diffuse & tufts papillae); 3 = Moderate (moderate & tufts papillae); 4 = Severe (giant papillae). The maximum of the four zones was selected for the analysis. Both eyes were included in the model for analysis. A higher change value indicates a larger reduction in the severity of the lid papillae.
Time Frame: Baseline (Day 0), Day 90
Population: This analysis group includes all subjects exposed to a study regimen with post baseline efficacy assessments. No imputation methods were employed; therefore only efficacy measurements available at each visit and time point were analyzed. Here, "n" is subjects with non-missing values at the specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Clear Care, Right Eye; Clear Care, Left Eye: Hydrogen peroxide-based contact lens solution used with habitual contact lenses for 90 days
- Habitual MPS, Right Eye; Habitual MPS, Left Eye: Habitual contact lens solution used with habitual contact lenses for 90 days
Arm/Group | Clear Care, Right Eye | Clear Care, Left Eye | Habitual MPS, Right Eye | Habitual MPS, Left Eye
Number analyzed (Participants) | 64 | 64 | 67 | 67
units on a scale
  Baseline (Day 0) | 2.3 (0.54) | 2.3 (0.62) | 2.2 (0.54) | 2.2 (0.54)
  Change from baseline at Day 90 (n=61, 61, 67, 67) | 0.9 (0.74) | 0.9 (0.81) | 0.5 (0.56) | 0.3 (0.69)

2. Secondary Outcome: Top 2 Box Percentage Agreement for "My Lenses Feel Like New" at Day 90
Description: As interpreted and reported by the subject on a questionnaire. A 5-point Likert scale was used, where 1=strongly disagree; 2=disagree; 3=undecided; 4=agree; 5=strongly agree. The Top-2-box response (agree, strongly agree) was calculated and reported as a percentage of all responses.
Time Frame: Day 90
Population: This analysis group includes all subjects exposed to a study regimen with post baseline efficacy assessments. No imputation methods were employed; therefore only efficacy measurements available at each visit and time point were analyzed.
Measure: Number; unit: percentage of subjects
Arm/Group | Clear Care | Habitual MPS
Number analyzed (Participants) | 61 | 67
percentage of subjects | 52.5 | 37.3

3. Secondary Outcome: Mean Frequency Score for Symptoms of Grittiness at Day 90
Description: As interpreted and reported by the subject on a questionnaire. The subject was asked, "During a typical day in the past 2 weeks, how often did your eyes feel gritty and/or scratchy while wearing your contact lenses?" and responded on a 5-point scale (1 = Never; 2 = Rarely; 3 = Sometimes; 4 = Frequently; 5 = Constantly).
Time Frame: Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clear Care | Habitual MPS
Number analyzed (Participants) | 61 | 67
units on a scale | 1.7 (0.90) | 2.3 (0.95)

4. Secondary Outcome: Mean Frequency Score for Symptoms of Dryness at Day 90
Description: As reported and interpreted by the subject on a questionnaire. The subject was asked "During a typical day in the past 2 weeks, how often did your eyes feel dry?" and responded on a 5-point scale ((0 = Never; 1 = Rarely; 2 = Sometimes; 3 = Frequently; 4 = Constantly).
Time Frame: Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clear Care | Habitual MPS
Number analyzed (Participants) | 61 | 67
units on a scale | 1.2 (0.87) | 1.8 (0.99)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (DEC 2013 - MAY 2014). This analysis group includes all subjects who were exposed to a study regimen.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device.
Arm/Group | Clear Care | Habitual MPS
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/68
Other Adverse Events (participants affected / at risk) | 0/66 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.